CLINICAL TRIAL: NCT01674803
Title: Comparison of BIOdegradable Polymer and DuRablE Polymer Drug-eluting Stents in an All COmeRs PopulaTion: Randomized Multicenter Trial in an All Comers Population Treated Within thE NeThErlands 3 (TWENTE 3)
Brief Title: Comparison of BIOdegradable Polymer and DuRablE Polymer Drug-eluting Stents in an All COmeRs PopulaTion (BIO-RESORT)
Acronym: BIO-RESORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation of Cardiovascular Research and Education Enschede (Other)
Responsible Party: Principal Investigator, prof. C. von Birgelen, Professor C. von Birgelen, Thorax Centrum Twente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIO-RESORT
Record Dates: First submitted 2012-08-21; First posted 2012-08-29 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Acute Coronary Syndrome; Angina Pectoris; Angina, Unstable; Myocardial Infarction; Coronary Artery Disease; Coronary Stenosis; Coronary Restenosis
Keywords: drug-eluting stent; zotarolimus; everolimus; sirolimus; all comers population; target vessel failure; coronary artery disease; durable polymer; biodegradable polymer
MeSH Terms: conditions — Acute Coronary Syndrome; Angina Pectoris; Angina, Unstable; Myocardial Infarction; Coronary Artery Disease; Coronary Stenosis; Coronary Restenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Orsiro (Active Comparator)
  Interventions: Device: Orsiro
- Synergy (Active Comparator)
  Interventions: Device: Synergy
- Resolute Integrity (Active Comparator)
  Interventions: Device: Resolute Integrity

INTERVENTIONS:
Device: Orsiro — biodegradable polymer sirolimus eluting stent
  Arms: Orsiro
Device: Synergy — biodegradable polymer everolimus eluting stent
  Arms: Synergy
Device: Resolute Integrity — durable polymer zotarolimus-eluting stent
  Arms: Resolute Integrity

SUMMARY:
The introduction of drug-eluting stents (DES) in the treatment of coronary artery disease has led to a significant reduction in morbidity. However, the first generation of these devices had no positive impact on the mortality after PCI (compared to bare metal stents), which was greatly attributed to a somewhat increased incidence of late and very late stent thrombosis. Concerns about the role of durable polymers as a potential trigger of inflammation and finally adverse events also led to the development of DES with biodegradable coatings, which leave after degradation of the coating only a bare metal stent in the vessel wall that does not induce an inflammatory response. While such biodegradable polymer DES are increasingly used in clinical practice, there is no data available from head-to-head comparisons between biodegradable and contemporary third generation durable polymer DES.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years.
* Significant coronary artery disease and lesion(s) eligible for treatment with drug eluting stents according to clinical guidelines and/or the operators' judgement.
* Capable of providing informed consent.
* Patients with all clinical syndromes will be enrolled without any exclusion based on number, type, location, or length of lesions to be treated.

Exclusion Criteria:

* Known intolerance to components of one of the stents that will be investigated or known intolerance to antithrombotic and/or anticoagulant therapy that prevents adherence to dual antiplatelet therapy.
* Planned elective surgical procedure necessitating interruption of dual antiplatelet therapy during the first 6 months after randomization.
* Participation in another randomized drug or device trial before reaching primary endpoint.
* Adherence to scheduled follow-up is unlikely or life expectancy assumed to be less than 1 year.
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3514 (Actual)
Dates: Start 2012-12-21 (Actual); Primary Completion 2016-08-24 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Target vessel failure (TVF) | 1 year
  Target vessel failure is a combined endpoint of cardiac death, target vessel related myocardial infarction and clinically driven target vessel revascularization.

SECONDARY OUTCOMES:
Target lesion failure (TLF) | 1 year
  Target lesion failure is a combined endpoint of cardiac death, target vessel related myocardial infarction, and clinically driven target lesion revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Albert Schweitzer Ziekenhuis, Dordrecht, Netherlands

REFERENCES:
- [Derived] Pinxterhuis TH, Ploumen EH, Zocca P, Doggen CJM, Schotborgh CE, Anthonio RL, Roguin A, Danse PW, Benit E, Aminian A, Hartmann M, Linssen GCM, von Birgelen C. Impact of premature coronary artery disease on adverse event risk following first percutaneous coronary intervention. Front Cardiovasc Med. 2023 Sep 7;10:1160201. doi: 10.3389/fcvm.2023.1160201. eCollection 2023. PMID 37745109
- [Derived] Pinxterhuis TH, Ploumen EH, Zocca P, Doggen CJM, Schotborgh CE, Anthonio RL, Roguin A, Danse PW, Benit E, Aminian A, van Houwelingen KG, Linssen GCM, Geelkerken RH, von Birgelen C. Outcome of percutaneous coronary intervention using ultrathin-strut biodegradable polymer sirolimus-eluting versus thin-strut durable polymer zotarolimus-eluting stents in patients with comorbid peripheral arterial disease: a post-hoc analysis from two randomized trials. Cardiovasc Diagn Ther. 2023 Aug 31;13(4):673-685. doi: 10.21037/cdt-22-584. Epub 2023 Jul 24. PMID 37675090
- [Derived] Pinxterhuis TH, Ploumen EH, Doggen CJM, Hartmann M, Schotborgh CE, Anthonio RL, Roguin A, Danse PW, Benit E, Aminian A, Linssen GCM, von Birgelen C. First myocardial infarction in patients with premature coronary artery disease: insights into patient characteristics and outcome after treatment with contemporary stents. Eur Heart J Acute Cardiovasc Care. 2023 Nov 16;12(11):774-781. doi: 10.1093/ehjacc/zuad098. PMID 37619976
- [Derived] Ploumen EH, Pinxterhuis TH, Buiten RA, Zocca P, Danse PW, Schotborgh CE, Scholte M, Gin RMTJ, Somi S, van Houwelingen KG, Stoel MG, de Man HAF, Hartmann M, Linssen GCM, van der Heijden LC, Kok MM, Doggen CJM, von Birgelen C. Final 5-Year Report of the Randomized BIO-RESORT Trial Comparing 3 Contemporary Drug-Eluting Stents in All-Comers. J Am Heart Assoc. 2022 Nov 15;11(22):e026041. doi: 10.1161/JAHA.122.026041. Epub 2022 Nov 8. PMID 36346050
- [Derived] Pinxterhuis TH, Ploumen EH, Zocca P, Doggen CJM, Schotborgh CE, Anthonio RL, Roguin A, Danse PW, Benit E, Aminian A, Stoel MG, Linssen GCM, Geelkerken RH, von Birgelen C. Outcome after percutaneous coronary intervention with contemporary stents in patients with concomitant peripheral arterial disease: A patient-level pooled analysis of four randomized trials. Atherosclerosis. 2022 Aug;355:52-59. doi: 10.1016/j.atherosclerosis.2022.05.002. Epub 2022 May 20. PMID 35641327
- [Derived] Ploumen EH, Pinxterhuis TH, Zocca P, Roguin A, Anthonio RL, Schotborgh CE, Benit E, Aminian A, Danse PW, Doggen CJM, von Birgelen C, Kok MM. Impact of prediabetes and diabetes on 3-year outcome of patients treated with new-generation drug-eluting stents in two large-scale randomized clinical trials. Cardiovasc Diabetol. 2021 Oct 30;20(1):217. doi: 10.1186/s12933-021-01405-4. PMID 34717627
- [Derived] Buiten RA, Ploumen EH, Zocca P, Doggen CJM, van Houwelingen KG, Danse PW, Schotborgh CE, Stoel MG, Scholte M, Linssen GCM, de Man FHAF, von Birgelen C. Three contemporary thin-strut drug-eluting stents implanted in severely calcified coronary lesions of participants in a randomized all-comers trial. Catheter Cardiovasc Interv. 2020 Nov;96(5):E508-E515. doi: 10.1002/ccd.28886. Epub 2020 Apr 1. PMID 32237060
- [Derived] Buiten RA, Ploumen EH, Zocca P, Doggen CJM, Danse PW, Schotborgh CE, Scholte M, van Houwelingen KG, Stoel MG, Hartmann M, Tjon Joe Gin RM, Somi S, Linssen GCM, Kok MM, von Birgelen C. Thin, Very Thin, or Ultrathin Strut Biodegradable or Durable Polymer-Coated Drug-Eluting Stents: 3-Year Outcomes of BIO-RESORT. JACC Cardiovasc Interv. 2019 Sep 9;12(17):1650-1660. doi: 10.1016/j.jcin.2019.04.054. Epub 2019 Aug 14. PMID 31422087
- [Derived] Buiten RA, Ploumen EH, Zocca P, Doggen CJM, van der Heijden LC, Kok MM, Danse PW, Schotborgh CE, Scholte M, de Man FHAF, Linssen GCM, von Birgelen C. Outcomes in Patients Treated With Thin-Strut, Very Thin-Strut, or Ultrathin-Strut Drug-Eluting Stents in Small Coronary Vessels: A Prespecified Analysis of the Randomized BIO-RESORT Trial. JAMA Cardiol. 2019 Jul 1;4(7):659-669. doi: 10.1001/jamacardio.2019.1776. PMID 31111862
- [Derived] von Birgelen C, Kok MM, van der Heijden LC, Danse PW, Schotborgh CE, Scholte M, Gin RMTJ, Somi S, van Houwelingen KG, Stoel MG, de Man FHAF, Louwerenburg JHW, Hartmann M, Zocca P, Linssen GCM, van der Palen J, Doggen CJM, Lowik MM. Very thin strut biodegradable polymer everolimus-eluting and sirolimus-eluting stents versus durable polymer zotarolimus-eluting stents in allcomers with coronary artery disease (BIO-RESORT): a three-arm, randomised, non-inferiority trial. Lancet. 2016 Nov 26;388(10060):2607-2617. doi: 10.1016/S0140-6736(16)31920-1. Epub 2016 Oct 30. PMID 27806902
- [Derived] Lam MK, Sen H, Tandjung K, van Houwelingen KG, de Vries AG, Danse PW, Schotborgh CE, Scholte M, Lowik MM, Linssen GC, Ijzerman MJ, van der Palen J, Doggen CJ, von Birgelen C. Comparison of 3 biodegradable polymer and durable polymer-based drug-eluting stents in all-comers (BIO-RESORT): rationale and study design of the randomized TWENTE III multicenter trial. Am Heart J. 2014 Apr;167(4):445-51. doi: 10.1016/j.ahj.2013.11.014. Epub 2014 Jan 6. PMID 24655691